CLINICAL TRIAL: NCT06783751
Title: Mechanistic and Clinical Outcomes of a Surgical Innovation Aimed at Minimizing GERD Associated With Vertical Sleeve Gastrectomy (INNOVATE-VSG)
Brief Title: Mechanistic and Clinical Outcomes of a Surgical Innovation Aimed at Minimizing GERD Associated With VSG (INNOVATE-VSG)
Acronym: INNOVATE-VSG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, San Diego (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Nihn Tuan Nguyen, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3451; 1R01DK138047-01A1 (NIH)
Record Dates: First submitted 2025-01-02; First posted 2025-01-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Bariatric Surgery; Sleeve Gastrectomy; Gastroesophageal Reflux Disease
MeSH Terms: conditions — Obesity; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Vertical Sleeve Gastrectomy (mVSG) (Experimental): modified investigational vertical sleeve gastrectomy (mVSG)
  Interventions: Procedure: Modified Vertical Sleeve Gastrectomy (mVSG)
- Conventional Vertical Sleeve Gastrectomy (cVSG) (Active Comparator): conventional vertical sleeve gastrectomy (cVSG)
  Interventions: Procedure: Conventional Vertical Sleeve Gastrectomy (cVSG)

INTERVENTIONS:
Procedure: Modified Vertical Sleeve Gastrectomy (mVSG) — The modified procedure preserves the gastric sling fibers and re-establishes the gastroesophageal flap valve (GEFV).
  Arms: Modified Vertical Sleeve Gastrectomy (mVSG)
Procedure: Conventional Vertical Sleeve Gastrectomy (cVSG) — Vertical Sleeve Gastrectomy as standard procedure
  Arms: Conventional Vertical Sleeve Gastrectomy (cVSG)

SUMMARY:
This is a two-site randomized clinical trial aiming to test whether a modified investigational bariatric surgical procedure can improve gastroesophageal reflux disease (GERD) after sleeve gastrectomy.

DETAILED DESCRIPTION:
The study will examine whether a modified vertical sleeve gastrectomy (mVSG) will improve GERD and quality of life.

Aim 1 (Primary): to determine whether mVSG, in comparison to conventional vertical sleeve gastrectomy (cVSG), will be associated with lower acid exposure time (AET, measured by the Bravo pH test) at 6-9 months. The investigators hypothesize that, at Month 6-9, compared to cVSG:

• H1. mVSG will be associated with lower AET

Aim 2 (Secondary): To elucidate the mechanistic basis for Aim 1, the investigators will perform following tests, before and at 6-9 months post-surgery: a) High resolution esophageal manometry (HREM) to determine the lower esophageal sphincter (LES) and intragastric pressure; b) The endoluminal functional lumen imaging probe (EndoFLIP) testing to examine changes in compliance of the LES; c) Measure the length of the gastroesophageal flap valve (GEFV) on the retroflex view during endoscopic exam. The investigators hypothesize that, at Month 6-9, compared to cVSG:

* H2a. mVSG will be associated with higher LES pressure and lower intragastric pressure
* H2b. mVSG will be associated with lower LES compliance
* H2c. GEFV will be present after mVSG (vs absence after cVSG)

Aim 3: Examine the impact of GERD on quality of life (QoL) with two validated rating scales - Gastroesophageal reflux disease-health related quality of life (GERD-HRQL) and Short Form-36 (SF-36). The investigators hypothesize that, at 12 months, compared to cVSG:

• H3. mVSG will lead to superior QoL

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18-65 years
2. Body mass index (BMI) 35-55 kg/m2
3. Must meet the BMI criteria before and after 6 months of nonsurgical weight management
4. Presence of GERD defined for this trial as acid exposure time (AET) of 4.9% or above as assessed with the Bravo pH test.
5. Have health insurance which pays for the costs of bariatric surgery and standard medical care before and after surgery
6. Women of childbearing potential must be using appropriate contraception to avoid pregnancy throughout the study, and must have a negative pregnancy test at study entry and prior to surgery
7. Must be able to provide written informed consent

Exclusion Criteria:

1. Hiatal hernia >2cm (defined as maximum axial height from end of the esophagus to diaphragm by any study including upper endoscopy esophagram and or at the time of surgery)
2. Evidence of clinically significant major esophageal motility disorder as determined by the site primary investigator
3. Severe gastroparesis
4. Previous bariatric or anti-reflux procedure
5. Barrett's esophagus
6. Subjects requiring mesh treatment at time of procedure
7. Severe heart (e.g., severe heart failure, unstable coronary artery disease), or end-stage lung disease as determined by the site primary investigator
8. Subjects with pacemakers, implantable defibrillators, neurostimulators
9. Portal hypertension or cirrhosis
10. Chronic pancreatitis
11. Active cancer treatment
12. Inability to tolerate general anesthesia
13. Uncontrollable coagulopathy
14. Significant and uncontrolled inflammatory bowel disease
15. Severe and/or uncontrolled psychiatric disorder (including psychosis, bipolar disorder) as determined during standard pre-surgery psychiatric screening at the site.
16. Suicidal ideation or unstable/untreated major depressive disorder within the past year
17. Alcohol or substance use disorder within the past year.
18. Pregnant or breastfeeding or planning pregnancy in the coming 24 months
19. Diminished intellectual capacity to consent or follow pre- and post-surgery instructions
20. History of, or any current health condition that, in the opinion of the PI, would make the subject ineligible for sleeve gastrectomy, or put the subject at risk by participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
% Acid Exposure Time (%AET) | Pre-surgery, Month 6-9 post surgery
  Change in %AET in percentage points at Month 6-9 relative to pre-surgery %AET assessed with the Bravo pH test

SECONDARY OUTCOMES:
LES pressure | Pre-surgery, Month 6-9 post surgery
  Change in LES pressure in millimeters of mercury (mmHg) assessed with High Resolution Esophageal Manometry (HREM)
Intragastric pressure | Pre-surgery, Month 6-9 post surgery
  Change in intragastric pressure in millimeters of mercury (mmHg) assessed with HREM
LES compliance | Pre-surgery, Month 6-9 post surgery
  Change in LES compliance in ratio of mm3/mmHg assessed with EndoFLIP
GEFV length | Pre-surgery, Month 6-9 post surgery
  Change in GEFV length in millimeters (mm) assessed with endoscopic exam

OTHER OUTCOMES:
GERD-HRQL score | Pre-surgery, Months 4, 6-9, 12 post surgery
  Change in GERD-HRQL score assessed with GERD-HRQL questionnaire
Health-related quality of life | Pre-surgery, Months 4, 6-9, 12 post surgery
  Change in SF-36 score assessed with SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ninh T. Nguyen, MD, Principal Investigator — University of California, Irvine; Ravinder K. Mittal, MD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California, Irvine, Orange, California
  - University of California, San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No